CLINICAL TRIAL: NCT07142044
Title: Safety, Tolerability and Exploratory Efficacy of EC5026 in Parkinson's Disease (STEP Study)
Acronym: STEP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EicOsis Human Health Inc. (Industry)
Collaborators: University of California, Davis (Other); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC5026-1-05
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease (PD)
Keywords: EC5026; Parkinson's Disease; Soluble Epoxide Hydrolase; sEH; Soluble Epoxide Hydrolase inhibitor
MeSH Terms: interventions — EC5026

STUDY DESIGN:
Intervention Model Description: This study will consist of two independent dose cohorts, Cohort 1 and Cohort 2. Each cohort will enroll eighteen (9) unique participants.
  In each cohort, 9 adults with Parkinson's Disease will be randomized to receive EC5026 or a matching placebo (2:1 randomization ratio). EC5026 and placebo will be administered orally in tablets, once daily, for 28 consecutive days. In Cohort 1, study participants will receive a daily dose of 2 mg of EC5026 or matching placebo; in Cohort 2, study participants will receive a daily dose of 4 mg of EC5026 or matching placebo. Dosing will be inpatient for the first 4 doses (facility discharge on Day 4 of the study period) and outpatient thereafter. There will be a 28 day follow up period after receiving the last dose of EC5026 or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EC5026 2 mg daily (Experimental): Once-daily, oral dose of 2 mg of EC5026 for 28 consecutive days
  Interventions: Drug: EC5026 oral tablet
- EC5026 4 mg daily (Experimental): Once-daily, oral dose of 4 mg of EC5026 for 28 consecutive days
  Interventions: Drug: EC5026 oral tablet
- Placebo (Placebo Comparator): Once-daily, matching placebo for each dose cohort, orally for 28 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EC5026 oral tablet — Oral soluble epoxide hydrolase inhibitor
  Arms: EC5026 2 mg daily; EC5026 4 mg daily
Drug: Placebo — Matching oral placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the oral drug candidate EC5026 is safe and targets the correct pathways to treat Parkinson's Disease in adults. It will also learn about the levels of drug that are achieved in blood and in the fluid surrounding the brain (spinal fluid). The main questions it aims to answer are:

* Is EC5026 safe in adults with Parkinson's Disease?
* What are the levels of EC5026 achieved after oral administration for 28 days?
* What molecules or pathways does EC5026 target, and to what extent?

In addition, although it is not one of the primary aims of the study, this clinical trial will also explore if oral administration of EC5026 improves the symptoms of Parkinson's Disease.

Researchers will compare EC5026 to a placebo (a look-alike substance that contains no drug).

Participants will:

* Take EC5026 or a placebo every day for 28 consecutive days
* Visit the clinic for frequent checkups, blood tests, spinal fluid tests, and questionnaires

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled Phase 1b multiple ascending dose (MAD) study to be conducted in adult male and female participants with Parkinson's Disease. The aim is to evaluate the safety, pharmacokinetics (PK), target engagement, and exploratory efficacy, of 2 ascending dose regimens of oral EC5026 in participants with Parkinson's Disease.

The study drug, EC5026, is an orally bioavailable inhibitor of an enzyme, soluble epoxide hydrolase (sEH), that is being developed as a first-in-class anti-inflammatory agent. Inhibiting sEH maintains concentrations of bioavailable polyunsaturated fatty acid epoxides, known as epoxy fatty acids (EpFAs). EpFAs are potent, endogenous fatty acids that are highly produced in areas of damaged and inflamed tissue but are rapidly metabolized by sEH in vivo. Therefore, selective inhibition of sEH prolongs and enhances the anti-inflammatory activity of EpFAs. Several studies have identified the sEH enzyme as a potential therapeutic target for modulating neuroinflammatory responses in PD.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females, 50 to 80 years of age (inclusive) at the time of Screening.
2. Able to understand the consent form, and to provide voluntary written informed consent.
3. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures to complete the study.
4. Confirmed diagnosis of idiopathic Parkinson's Disease according to 2015 Movement Disorder Society (MDS) clinical diagnostic criteria.
5. Off state Hoehn & Yahr below Stage 3 at the time of Screening.
6. Participants must be on stable doses of L-dopa with or without other adjunctive PD therapy for at least 30 days prior to enrollment. Doses should be expected to remain stable for the duration of the study.
7. Participants must be in overall stable condition, as determined by pre-study medical history, physical examination, clinical laboratory tests, and 12 lead ECG measurements.
8. Participants must have normal or not clinically significant clinical laboratory test results, as determined by the study investigator, including coagulation panel, blood cell counts, comprehensive metabolic panel analytes, and creatinine clearance (60 cm3/min or greater). Clinical laboratory tests results that are consistent with known, stable comorbidities will be allowed as long as the comorbidities do not represent an exclusion criteria per se.
9. Participants must have a negative urinary drug screen (UDS) for illicit drugs and a negative alcohol breath test.
10. Abstention from use of other investigative or non-approved drugs for the duration of the trial
11. Male participants who are not surgically sterile (vasectomized) and their female sexual partners must agree to use contraception during the study period and for 2 months after receiving the last dose of study drug.
12. Male participants must not donate sperm during the study and for 12 months after receiving the last dose of study drug.
13. Female participants must be non-pregnant, non-lactating, and either postmenopausal for at least 1 year, or surgically sterile (bilateral tubal ligation, 'clipping or tying tubes,' or hysterectomy) for at least 3 months, or they must agree to use two forms of highly effective contraception method (less than 1 pregnancy per 100 people using the method for one year) from 28 days and/or their last confirmed menstrual period prior to study enrollment (whichever is longer) until 2 months after receiving the last dose of study drug. Postmenopausal status will be defined as follows: minimum 1 year; amenorrhea duration of 12 consecutive months and a serum FSH value >40 IU/L; postmenopausal status must be confirmed by an FSH test at Screening). Highly effective contraception methods include: Intra-uterine device (IUD) containing either copper or levonorgestrel (e.g., Mirena®), and/or barrier methods of contraception, including condoms (external or internal) and diaphragm ('cap'). Hormonal methods of contraception (with the exception of hormonal IUD) are not permitted within this study. Female participants will refrain from using hormonal contraceptives for at least 28 days prior to study entry until the end of the study period. Participants/Participant's partner(s) must also use a barrier form of contraception, from the first dose of study drug through until 2 months after the last dose. For all females of childbearing potential, the pregnancy test result must be negative at Screening and Pre-Study Baseline (Day -1).
14. Participants must be able to speak, read, and understand English sufficiently to allow comprehension and completion of all study assessments.

Exclusion Criteria:

1. Atypical parkinsonian syndrome or secondary parkinsonism (e.g., due to drugs or toxins, metabolic neurogenetic disorders, encephalitis, cerebrovascular disease or non-PD degenerative disease).
2. Family history of early onset PD (age <50 years) or known personal genetically causal etiology of PD.
3. Diagnosis of any other clinically significant neurologic disease that may confound the assessment of the study drug on PD symptoms
4. Not stabilized with current therapeutic regimen for PD or likely to require changes in L-dopa therapy over the duration of the trial.
5. Presence of PD psychosis or dementia, or other neuropsychiatric or psychiatric conditions impeding informed consent or compliance with study interventions.
6. Severe dyskinesia (defined as per MDS-UPDRS) during a "normal day" that would significantly interfere with the participant's ability to perform study assessments.
7. History of neurosurgery for PD or tremor.
8. Clinically significant medical, surgical, or laboratory abnormalities in the judgement of the Investigator.
9. Participants with any clinically unstable or significant cardiovascular (including acute coronary syndrome within the prior year to Screening), renal, hepatic, respiratory, gastrointestinal, hematological, endocrine, or infectious disease (including HIV infection).
10. Participants with clinically significant abnormalities on screening vital signs, laboratory tests, and/or ECG, per investigator's judgement. Participants with poor venous access will also be excluded.
11. Participants with a family history of significant cardiac disease (i.e., sudden death in first degree relative; myocardial infarction before the age of 50).
12. Participants with a history of disorders of the hypothalamic-pituitary-adrenal axis, including adrenal insufficiency and Cushing's, or with a history of disorders of the hypothalamic-pituitary-gonadal axis, including hypogonadism.
13. Participants with any of the following blood values at screening:

    * Abnormal plasma renin and/or aldosterone value
    * Morning cortisol level <5 mcg/dL
    * ACTH stimulated cortisol levels <18 mcg/dL at 60 minutes after ACTH injection at screening, or
    * Abnormal FSH, LH, testosterone (for males), or estradiol (for females, unless post-menopausal)
14. Participants who have used any topical, oral, or intravenous exogenous corticosteroids within 12 weeks and/or intra-articular exogenous corticosteroids within 6 months prior to the start of the trial, or who plan on using them during the study.
15. Participants who have used chemotherapy agents, or who have a personal history of cancer or cancer in first degree relatives suggestive of elevated cancer risk, other than nonmetastatic skin cancer that has been completely excised, within 5 years prior to Screening.
16. Participants who have used (within 14 days of randomization) or plan on using during the duration of the study any prescription or over-the-counter drugs that are moderate or strong CYP3A4 inducers or inhibitors.
17. Participants who have used (within 14 days of randomization) or plan on using during the duration of the study any dietary aids, supplements, or foods that are moderate or strong CYP3A4 inhibitors (e.g., grapefruit juice).
18. Participants with difficulty in swallowing oral medications
19. Participants who have used any other investigational drug within 1 month or 5 half-lives, whichever is longer, prior to enrollment.
20. Participants with a documented history of difficult lumbar puncture procedures, to the investigator's discretion.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAE) [Safety and Tolerability] | 56 days
  All AEs reported or observed during the study will be recorded on the electronic case report forms (eCRF). Information to be collected includes drug treatment, type of event, time of onset, dosage, investigator-specified assessment of severity and relationship to study drug, time of resolution of the event, seriousness, any required treatment or evaluations, and outcome. Any AEs resulting from concurrent illnesses, reactions to concurrent illnesses, reactions to concurrent medications, or progression of disease states must also be reported. All AEs will be followed until they are resolved, stable, or judged by the investigator to be not clinically significant. The Medical Dictionary for Regulatory Activities will be used to code all AEs.

OTHER OUTCOMES:
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on plasma and cerebrospinal fluid levels of EC5026 | 56 days
  Standard validated EC5026 measurement platform will be used
Effects of 2 ascending multiple dose regimens of EC5026 versus placebo on plasma and cerebrospinal fluid target engagement biomarkers. | 56 days.
  Target engagement biomarkers will include changes from baseline of a validated analytical platform of inflammatory cytokines, neurological markers including target inflammatory genes tied to the mechanism of action, ER-stress response genes, and Parkinson's Disease specific biomarkers (including alpha-synuclein, Abeta42, pTau-181, GFAP, and Neurofilament Light).
Change from Baseline in Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Score (Day 14) | Day 14
  Change from Baseline in Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Score on Day 14.
  The Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) is a comprehensive tool used to assess Parkinson's Disease (PD) symptoms and severity through a series of questions rated by clinicians, patients, and caregivers. Scores are on a 0-4 scale, with higher scores indicating a greater impact of PD symptoms. The scale is divided into four parts, covering non-motor and motor experiences of daily living, motor examination, and motor complications.
Change from Baseline in Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Score (Day 28) | Day 28
  Change from Baseline in Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Score on Day 28.
  The Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) is a comprehensive tool used to assess Parkinson's Disease (PD) symptoms and severity through a series of questions rated by clinicians, patients, and caregivers. Scores are on a 0-4 scale, with higher scores indicating a greater impact of PD symptoms. The scale is divided into four parts, covering non-motor and motor experiences of daily living, motor examination, and motor complications.
Change from Baseline in Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Score (Day 56 - End of Study) | Day 56
  Change from Baseline in Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) Score on Day 56 or end of study visit.
  The Movement Disorders Society-Unified Parkinson Disease Rating Scale (MDS-UPDRS) is a comprehensive tool used to assess Parkinson's Disease (PD) symptoms and severity through a series of questions rated by clinicians, patients, and caregivers. Scores are on a 0-4 scale, with higher scores indicating a greater impact of PD symptoms. The scale is divided into four parts, covering non-motor and motor experiences of daily living, motor examination, and motor complications.
Change from Baseline in Movement Disorders Society Non-Motor Symptom Scale (NMS) (Day 14) | Day 14
  Change from Baseline in Movement Disorders Society Non-Motor Symptom Scale (NMS) on Day 14.
  The Movement Disorders Society (MDS) Non-Motor Symptom Scale (MDS-NMS) is evaluates 52 items, grouped according to clinical content into 13 domains. Items are scored for frequency (from 0 [never] to 4 [majority of time]) and severity (from 0 [not present] to 4 [severe]), which are multiplied to generate the item total score. Scores for each domain and the total rating scale (maximum, 832 points) are calculated by summing the corresponding items. The scale provides a total score representing the non-motor burden. Higher scores imply a higher non-motor symptom burden.
Change from Baseline in Movement Disorders Society Non-Motor Symptom Scale (NMS) (Day 28) | Day 28
  Change from Baseline in Movement Disorders Society Non-Motor Symptom Scale (NMS) on Day 28.
  The Movement Disorders Society (MDS) Non-Motor Symptom Scale (MDS-NMS) is evaluates 52 items, grouped according to clinical content into 13 domains. Items are scored for frequency (from 0 [never] to 4 [majority of time]) and severity (from 0 [not present] to 4 [severe]), which are multiplied to generate the item total score. Scores for each domain and the total rating scale (maximum, 832 points) are calculated by summing the corresponding items. The scale provides a total score representing the non-motor burden. Higher scores imply a higher non-motor symptom burden.
Change from Baseline in Movement Disorders Society Non-Motor Symptom Scale (NMS) (Day 56 - End of Study) | Day 56
  Change from Baseline in Movement Disorders Society Non-Motor Symptom Scale (NMS) on Day 56 or end of study visit.
  The Movement Disorders Society (MDS) Non-Motor Symptom Scale (MDS-NMS) is evaluates 52 items, grouped according to clinical content into 13 domains. Items are scored for frequency (from 0 [never] to 4 [majority of time]) and severity (from 0 [not present] to 4 [severe]), which are multiplied to generate the item total score. Scores for each domain and the total rating scale (maximum, 832 points) are calculated by summing the corresponding items. The scale provides a total score representing the non-motor burden. Higher scores imply a higher non-motor symptom burden.
Change from Baseline in Time to Complete Time Up and Go (TUG) Test (Day 14) | Day 14
  Change from Baseline in Time to Complete Time Up and Go (TUG) Test on Day 14. The Time Up and Go (TUG) test time varies, but healthy older adults typically complete it in under 10 seconds. A score of 12 seconds or more indicates increased fall risk, with a threshold of 13.5 seconds often used for community-dwelling adults. Scores of 20 seconds or more signal poor physical performance and higher fall risk, while very frail individuals might take two minutes or more to finish.
Change from Baseline in Time to Complete Time Up and Go (TUG) Test (Day 28) | Day 28
  Change from Baseline in Time to Complete Time Up and Go (TUG) Test on Day 28. The Time Up and Go (TUG) test time varies, but healthy older adults typically complete it in under 10 seconds. A score of 12 seconds or more indicates increased fall risk, with a threshold of 13.5 seconds often used for community-dwelling adults. Scores of 20 seconds or more signal poor physical performance and higher fall risk, while very frail individuals might take two minutes or more to finish.
Change from Baseline in Time to Complete Time Up and Go (TUG) Test (Day 56 - End of Study) | Day 56
  Change from Baseline in Time to Complete Time Up and Go (TUG) Test on Day 56 or end of study visit.
  The Time Up and Go (TUG) test time varies, but healthy older adults typically complete it in under 10 seconds. A score of 12 seconds or more indicates increased fall risk, with a threshold of 13.5 seconds often used for community-dwelling adults. Scores of 20 seconds or more signal poor physical performance and higher fall risk, while very frail individuals might take two minutes or more to finish.
Change from Baseline in Clinical Global Impression (CGI) Scale (Day 14) | Day 14
  Change from Baseline in Clinical Global Impression (CGI) Scale on Day 14. The CGI was developed for use in NIMH-sponsored clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI has two components-the CGI-Severity, which rates illness severity (on a scale from 1 to 7), and the CGI-Improvement, which rates change from the initiation (baseline) of treatment (on a similar 7-point scale). Higher scores in the 7-point scale for each of the components implies worse severity (CGI-S) or a change to worse from baseline (CGI-I).
Change from Baseline in Clinical Global Impression (CGI) Scale (Day 28) | Day 28
  Change from Baseline in Clinical Global Impression (CGI) Scale on Day 28. The CGI was developed for use in NIMH-sponsored clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI has two components-the CGI-Severity, which rates illness severity (on a scale from 1 to 7), and the CGI-Improvement, which rates change from the initiation (baseline) of treatment (on a similar 7-point scale). Higher scores in the 7-point scale for each of the components implies worse severity (CGI-S) or a change to worse from baseline (CGI-I).
Change from Baseline in Clinical Global Impression (CGI) Scale (Day 56 - End of Study) | Day 56
  Change from Baseline in Clinical Global Impression (CGI) Scale on Day 56. The CGI was developed for use in NIMH-sponsored clinical trials to provide a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI has two components-the CGI-Severity, which rates illness severity (on a scale from 1 to 7), and the CGI-Improvement, which rates change from the initiation (baseline) of treatment (on a similar 7-point scale). Higher scores in the 7-point scale for each of the components implies worse severity (CGI-S) or a change to worse from baseline (CGI-I).
Change from Baseline in Parkinson's Disease Questionnaire (PDQ-39) total score (Day 14) | Day 14
  Change from Baseline in Parkinson's Disease Questionnaire (PDQ-39) total score on Day 14.
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month. Specifically, it assesses how often patients experience difficulties across the 8 quality of life dimensions of functioning and well-being. It uses a 5-point scale for each of the 39 questions as follows: 0 = Never; 1 = Rarely; 2 = Sometimes; 3 = Often; and 4 = Always. The minimum score is 0 that means good health, while the maximum score is 100 that is bad health; a higher score indicates a lower quality of life.
Change from Baseline in Parkinson's Disease Questionnaire (PDQ-39) total score (Day 28) | Day 28
  Change from Baseline in Parkinson's Disease Questionnaire (PDQ-39) total score on Day 28.
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month. Specifically, it assesses how often patients experience difficulties across the 8 quality of life dimensions of functioning and well-being. It uses a 5-point scale for each of the 39 questions as follows: 0 = Never; 1 = Rarely; 2 = Sometimes; 3 = Often; and 4 = Always. The minimum score is 0 that means good health, while the maximum score is 100 that is bad health; a higher score indicates a lower quality of life.
Change from Baseline in Parkinson's Disease Questionnaire (PDQ-39) total score (Day 56 - End of Study) | Day 56
  Change from Baseline in Parkinson's Disease Questionnaire (PDQ-39) total score on Day 56.
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month. Specifically, it assesses how often patients experience difficulties across the 8 quality of life dimensions of functioning and well-being. It uses a 5-point scale for each of the 39 questions as follows: 0 = Never; 1 = Rarely; 2 = Sometimes; 3 = Often; and 4 = Always. The minimum score is 0 that means good health, while the maximum score is 100 that is bad health; a higher score indicates a lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: William K Schmidt, PhD, Study Director — EicOsis Human Health Inc.; Lin Zhang, MD, PhD, Principal Investigator — UC Davis Health
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No